CLINICAL TRIAL: NCT06098664
Title: Observational Study of Sinus Rhythm Mapping in Pulmonary Vein Isolation Naive Patients With Atrial Fibrillation
Acronym: SUSTAINER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Laurent Pison, Clinical professor, Ziekenhuis Oost-Limburg
Other Study IDs: Z-2023039
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Artificial Intelligence; Deep Neural Network; Electrocardiogram; Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low score group (DNN-score = 0 - 10%): The inclusions will be stratified to the deep neural network (DNN) score. The study will enrol 20 patients in each group.
  Interventions: Diagnostic Test: AI-enabled ECG score for Atrial Fibrillation (DNN score); Diagnostic Test: Atrial voltage map in sinus rhythm
- Medium score group (DNN-score = 10 - 50%): The inclusions will be stratified to the deep neural network (DNN) score. The study will enrol 20 patients in each group.
  Interventions: Diagnostic Test: AI-enabled ECG score for Atrial Fibrillation (DNN score); Diagnostic Test: Atrial voltage map in sinus rhythm
- High score group (DNN-score = 50 - 100%): The inclusions will be stratified to the deep neural network (DNN) score. The study will enrol 20 patients in each group.
  Interventions: Diagnostic Test: AI-enabled ECG score for Atrial Fibrillation (DNN score); Diagnostic Test: Atrial voltage map in sinus rhythm

INTERVENTIONS:
Diagnostic Test: AI-enabled ECG score for Atrial Fibrillation (DNN score) — A 12-lead ECG, performed within 24 hours before the Pulmonary Vein Isolation (PVI) procedure, will be used to calculate the DNN score.
  (DNN score details: https://doi.org/10.1016/j.jacep.2023.04.008)
Diagnostic Test: Atrial voltage map in sinus rhythm — An atrial voltage map will be constructed prior to the PVI procedure.

SUMMARY:
Atrial fibrillation (AF) initially starts in a paroxysmal form, which is mainly based on the presence of triggers. Progression of AF is accompanied by structural and electrical remodelling which can typically be described as a progressive change in electrophysiological properties of the myocardium caused by cardiovascular comorbidities and AF itself. This results in complex electrical conduction disorders, which is defined as electropathology. The aim of our study is to evaluate whether an artificial intelligence (AI)-enabled ECG algorithm (on an ECG in Sinus Rhythm) can predict electropathology in patients with AF who undergo a first PVI.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent.
* First PVI-procedure
* Age is 18 years or higher.
* 12-lead ECG available in SR during the last 14 days.

Exclusion Criteria:

* Mitral insufficiency of grade 3 or 4.
* Participating in another study that may interfere with participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for a PVI will be consecutively screened and enrolled in the study. The inclusions will be stratified to the DNN score.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Low voltage area | During atrial voltage mapping, prior to PVI procedure.
  Proportion of low voltage area in the left atrium. (Defined as a threshold 0.5mV)

SECONDARY OUTCOMES:
Transition zone voltage area | During atrial voltage mapping, prior to PVI procedure.
  Proportion of transition zone voltage area in the left atrium. (Defined as a threshold 1mV)
Conduction delay | During atrial voltage mapping, prior to PVI procedure.
  Number of deceleration zones in the left atrium. (Deceleration zone defined as a zone with a conduction speed of <27cm/s)
Conduction delay score | During atrial voltage mapping, prior to PVI procedure.
  Weighted score for conduction deceleration zones (taking in account the number of affected zones and the severity of conduction delay)
Conduction time from sinus node to Bachman bundle | During atrial voltage mapping, prior to PVI procedure.
  Based on Local Activation Time (LAT) sampling. Defined as first point in right atrium to first point in left atrium.
Total LA conduction time | During atrial voltage mapping, prior to PVI procedure.
  Based on LAT sampling
Left atrial appendage ejection velocity. | Immediately prior to PVI procedure.
  Measured with TEE pulsed wave doppler.
Left atrial size | Prior to PVI procedure.
  Measured on CT or MRI imaging
Pericardial adipose tissue volume | Prior to PVI procedure.
  Measured on CT or MRI imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No